CLINICAL TRIAL: NCT06427811
Title: A Prospective, Multicenter, Single-arm, Open-label, Phase IV, Post-authorization Interventional Study to Assess the Safety and Efficacy of Asciminib in Indian Patients With Ph+ CML-CP (Without T315I Mutation), Previously Treated With Two or More Tyrosine Kinase Inhibitors and Ph+ CML-CP With T315I Mutation
Brief Title: Clinical Study of Asciminib in Previously Treated Indian Patients With Ph+ CML-CP Without T315I Mutation and in Patients With Ph+ CML-CP With T315I Mutation
Acronym: ASC4INDIA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABL001A2005
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Philadelphia Chromosome-Positive Chronic Myeloid Leukemia in Chronic Phase
Keywords: ABL001; Asciminib; Ph+ CML-CP; T315I mutation; Ph+ CML-CP without T315I mutation; Ph+ CML-CP with the T315I mutation; Myelogenous; Chronic; Chronic Myeloid Leukemia; Ph1 Positive Myeloid Leukemia; Philadelphia Positive Myeloid Leukemia; BCR-ABL Positive; Post-authorization Interventional Study; Tyrosine Kinase Inhibitors; TKI; Chronic Leukemia; Ph1 Positive Leukemia; Without T315I mutation; with the T315I mutation
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asciminib (Experimental): Participants without T315I mutation will receive 80 mg once daily at approximately the same time each day OR 40 mg twice daily per Investigator's discretion at approximately 12-hour intervals.
  Participants with T315I mutation will receive200 mg twice daily at approximately 12-hour intervals.
  Interventions: Drug: Asciminib

INTERVENTIONS:
Drug: Asciminib — Film-coated tablets with 40 mg dose strength taken orally
  Other Names: ABL001

SUMMARY:
The Drugs Controller General of India (DCGI) has granted approval for Asciminib film-coated 40 mg tablets on 20 Oct 2023 with the condition to perform a Phase IV clinical study in Indian patients with Philadelphia chromosome-positive chronic myeloid leukemia in chronic phase (Ph+ CML-CP) per the India Prescribing Information (PI). The purpose of this prospective, multicenter, single-arm, open-label, Phase IV study is, therefore, to confirm the safety and efficacy of Asciminib in Indian patients with Ph+ CML-CP (without threonine-315 residue with isoleucine [T315I] mutation), previously treated with 2 or more tyrosine kinase inhibitors (TKIs) and patients with Ph+ CML-CP with T315I mutation.

DETAILED DESCRIPTION:
This is a Phase IV, prospective, multicenter, single-arm, open-label, post-authorization interventional study to assess the safety and efficacy of asciminib in Indian participants with Ph+ CML-CP (without T315I mutation), previously treated with 2 or more TKIs and participants with Ph+ CML-CP with T315I mutation irrespective of the line of treatment.

The study will include 3 periods: a screening period (up to 21 days), a treatment period of up to 6 months with asciminib (with dosing according to mutation status), and a safety follow-up period for 30 days after the last dose of the study treatment. Completion of the safety follow-up period after the last dose of the study treatment will be considered as the End of Study (EOS).

After obtaining the written informed consent form (ICF) from the participant or their legally authorized representatives (LARs), the participants will undergo screening procedures to confirm their eligibility for the study.

The results of the breakpoint cluster region gene-Abelson proto-oncogene 1, nonreceptor tyrosine kinase gene (BCR::ABL1) real-time quantitative polymerase chain reaction (RQ-PCR) as well as the T315I mutation report need to be established and documented prior to enrollment into the study in the screening period in line with the inclusion criteria of the study. Participants with previously documented T315I mutated CML-CP will be directly considered for the screening procedures. If the status of the T315I mutation is not known, the participant will undergo a standardized Sanger sequencing/PCR/next-generation sequencing (NGS)-based T315I mutation test (as per the availability at the site).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male or female participants ≥18 years of age at the screening visit with a confirmed diagnosis of Ph+ CML-CP.

Participants must meet all of the following laboratory values as confirmed by the available reports of the peripheral blood test or bone marrow examination (performed within 12 months before the screening) at the screening visit to meet the criteria of Ph+ CML-CP:

* <15% blasts in peripheral blood and/or bone marrow
* <30% blasts plus promyelocytes in peripheral blood and/or bone marrow
* <20% basophils in the peripheral blood
* ≥50 x 109/L (≥50,000/mm3) platelets#
* No evidence of extramedullary leukemic involvement, apart from hepatosplenomegaly.

  #Transient prior therapy related thrombocytopenia (<50,000/mm3 for ≤30 days prior to screening) is acceptable.

  - a. For Ph+ CML-CP participants with T315I mutation, mutational analysis testing at any time point showing a documented T315I mutation.

  b. For Ph+ CML-CP participants without T315I mutation, at least 2 prior ATP-site TKIs (i.e., imatinib, nilotinib, bosutinib, dasatinib, or ponatinib) with failure* (adapted from the 2020 European LeukemiaNet [ELN] Recommendations) or intolerance** to the most recent TKI therapy at the time of screening.

  *Failure for Ph+ CML-CP participants (CP at the time of initiation of last therapy) is defined as meeting at least one of the following criteria:
* Three months after the initiation of therapy: >10% BCR::ABL1 on IS if confirmed within 1-3 months
* Six months after the initiation of therapy: BCR::ABL1 ratio >10% IS
* Twelve months after initiation of therapy: BCR::ABL1 ratio >1% IS
* At any time after the initiation of therapy, loss of CHR, MR2
* At any time after the initiation of therapy, the development of new BCR::ABL1 mutations which potentially cause resistance to current treatment
* At any time 12 months after the initiation of therapy, BCR::ABL1 ratio ≥1% IS or loss of MMR
* At any time after the initiation of therapy, new clonal chromosome abnormalities in Ph+ cells (CCA/Ph+)

  **Intolerance is defined as:
* Non-hematologic toxicity: Participants with grade .3 or 4 toxicity while on therapy, or with persistent grade 2 toxicity, unresponsive to optimal management,including dose adjustments (unless dose reduction is not considered in the best interest of the participant if the response is already suboptimal)
* Hematologic toxicity: Participants with grade 3 or 4 toxicity (absolute neutrophil count [ANC] or platelets) while on therapy that is recurrent after dose reduction to the lowest doses recommended by India PI.

  * ECOG performance status of 0, 1, or 2.
  * Evidence of typical BCR::ABL1 transcript (e14a2 and/or e13a2) at the time of screening which is amenable to standardized RQ-PCR quantification.
  * Participants must have adequate end organ function as per the investigator's judgement.
  * Participants must have the following electrolyte values within normal limits or corrected to be within normal limits with supplements prior to the first dose of study treatment:
* Potassium (potassium increase of up to 6.0 mmol/L is acceptable at study entry if associated with creatinine clearance within normal limits)
* Total calcium (corrected for serum albumin); (calcium increase of up to 12.5 mg/dL or 3.1 mmol/L is acceptable at study entry if associated with creatinine clearance within normal limits)
* Magnesium, except for magnesium increase >upper level of normal (ULN) - 3.0 mg/dL or >ULN - 1.23 mmol/L associated with creatinine clearance (calculated using Cockcroft-Gault formula) within normal limits.

Exclusion Criteria:

* Known second chronic phase of CML after previous progression to CML-AP/CML-BC.
* Previous treatment with a hematopoietic stem-cell transplantation.
* Cardiac or cardiac repolarization abnormality, including any of the following:

  * History within 6 months prior to starting study treatment of myocardial infarction (MI), angina pectoris, and coronary artery bypass graft (CABG)
  * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block (e.g., bifascicular block, Mobitz type II and third-degree AV block)
  * QT corrected for heart rate by Fridericia's cube root formula (QTcF) at screening ≥450 msec (both male and female participants)
  * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
* Risk factors for Torsades de Pointes (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
* Inability to determine the QTcF interval.1. Known second chronic phase of CML after previous progression to CML-AP/CML-BC.
* Previous treatment with a hematopoietic stem-cell transplantation.
* Cardiac or cardiac repolarization abnormality, including any of the following:

  * History within 6 months prior to starting study treatment of myocardial infarction (MI), angina pectoris, and coronary artery bypass graft (CABG)
  * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block (e.g., bifascicular block, Mobitz type II and third-degree AV block)
  * QT corrected for heart rate by Fridericia's cube root formula (QTcF) at screening ≥450 msec (both male and female participants)
  * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
* Risk factors for Torsades de Pointes (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
* Inability to determine the QTcF interval
* Concomitant medication(s) with a "Known risk of TdP" (per www.crediblemeds.org) that cannot be discontinued or replaced 7 days prior to starting study treatment by safe alternative medication.
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g., uncontrolled diabetes, active or uncontrolled infection, pulmonary hypertension).
* History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis.
* Known infection with human immunodeficiency virus (HIV) or active hepatitis B or C.
* Known presence of significant congenital or acquired bleeding disorder unrelated to cancer.
* History of other active malignancy within 3 years prior to study entry with the exception of previous or concomitant basal cell skin cancer and previous carcinoma in situ treated curatively.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery).
* Previous treatment with or known/suspected hypersensitivity to asciminib or any of its excipients.
* Participants must avoid consumption of grapefruit, Seville oranges, or products containing the juice of each during the entire study and 7 days before the first dose of study treatment, due to potential CYP3A4 interaction with the study treatment. Orange juice is allowed. Participants must avoid consumption of over-the-counter medications or herbal supplements as these can interact with each other and may alter the effects of asciminib.
* Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.
* Pregnant or breastfeeding women.
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant unless they are using highly effective methods of contraception.

Highly effective contraception methods include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Note that periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy (with or without hysterectomy) total hysterectomy or bilateral tubal ligation at least 6 weeks before taking study treatment). In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
* Male sterilization (vasectomy) of the male partner(s) of the female participant at least 6 months prior to screening. The vasectomized male partner should be the sole partner for that participant.
* Use of oral, injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example, hormone vaginal ring or transdermal hormone contraception. In the case of the use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
* Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age-appropriate history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least 6 weeks before taking study treatment. In the case of oophorectomy alone, women are considered menopausal and not of childbearing potential only when the reproductive status of the woman has been confirmed by a follow-up hormone level assessment.

  - If a participant is presenting with symptoms suggestive of possible Coronavirus Disease (COVID-19) infection, advise ruling it out by appropriate testing recommended by health authorities.
* Nucleic acid amplification tests for viral RNA (polymerase chain reaction), to measure current infection with SARS-CoV-2
* Antigen tests for rapid detection of SARS-CoV-2
* Antibody (serology) tests to detect the presence of antibodies to SARS-CoV-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events(AEs)/serious AEs (SAEs) in participants with Ph+ CML-CP without T315I mutation | up to 6 months
  Frequency and severity of adverse events(AEs)/serious AEs (SAEs) in participants with Ph+ CML-CP (without T315I mutation), previously treated with 2 or more TKIs up to 6 months
Frequency and severity of AEs/SAEs in participants with Ph+ CML-CP with T315I mutation | up to 6 months
  Frequency and severity of AEs/SAEs in participants with Ph+ CML-CP with T315I mutation up to 6 months

SECONDARY OUTCOMES:
Percentage of participants with dose interruptions, reductions, and discontinuation (without T3151 mutation) | up to 6 months
  Percentage of participants with dose interruptions, reductions, and discontinuation up to 6 months.
Percentage of participants achieving a complete hematologic response (CHR) at 3 and 6 months (without T3151 mutation) | 3 months, 6 months
  A CHR is defined as the presence of all of the following for ≥4 weeks: white blood count (WBC) <10 x 109/L, platelet count <450 x 109/L, basophils <5%, no blasts and promyelocytes in peripheral blood, myelocytes + metamyelocytes <5% in peripheral blood, no evidence of extramedullary disease, including spleen and liver.
Percentage of participants achieving early molecular response (EMR) at 3 and 6 months (without T3151 mutation) | 3 months, 6 months
  Levels of BCR::ABL1 transcripts will be determined by RQ-PCR testing of peripheral blood and analyzed at a central testing laboratory. Log reduction in BCR::ABL1 transcripts levels from the standardized baseline value, or the percent ratio of BCR::ABL1 transcripts versus control gene (ABL1) transcripts converted to a reference standard, will be calculated for each sample.
  Early molecular response (EMR) is defined as ≤10% BCR::ABL1 international scale (IS).
Percentage of participants achieving molecular response (MR2) at 3 and 6 months (without T3151 mutation) | 3 months, 6 months
  Levels of BCR::ABL1 transcripts will be determined by RQ-PCR testing of peripheral blood and analyzed at a central testing laboratory. Log reduction in BCR::ABL1 transcripts levels from the standardized baseline value, or the percent ratio of BCR::ABL1 transcripts versus control gene (ABL1) transcripts converted to a reference standard, will be calculated for each sample. The rate of MR2 is defined as ≥2 log reduction of BCR::ABL (transcript from standardized baseline or ≤1% BCR::ABL/ABL1 % by IS), measured by RQ-PCR.
Percentage of participants achieving major molecular response (MMR) at 3 and 6 months (without T3151 mutation) | 3 months, 6 months
  Levels of BCR::ABL1 transcripts will be determined by RQ-PCR testing of peripheral blood and analyzed at a central testing laboratory. Log reduction in BCR::ABL1 transcripts levels from the standardized baseline value, or the percent ratio of BCR::ABL1 transcripts versus control gene (ABL1) transcripts converted to a reference standard, will be calculated for each sample. Major molecular response (MMR) is defined as ≤0.1% BCR::ABL1 on the IS.
Percentage of participants achieving molecular response of MR4 and MR4.5 at 3 and 6 months of the treatment period (without T3151 mutation) | 3 months, 6 months
  Levels of BCR::ABL1 transcripts will be determined by RQ-PCR testing of peripheral blood and analyzed at a central testing laboratory. Log reduction in BCR::ABL1 transcripts levels from the standardized baseline value, or the percent ratio of BCR::ABL1 transcripts versus control gene (ABL1) transcripts converted to a reference standard, will be calculated for each sample.
  MR4 is defined ≤0.01% BCR::ABL1 on the IS. MR4.5 is defined as ≤0.0032% BCR::ABL1 on the IS.
Time to achieve complete hematologic response (without T3151 mutation) | up to 6 months
  Time to achieve a response level (hematologic or molecular) is defined as the time from the date of the first dose of study treatment to the first documented achievement of each defined response level. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Time to achieve early molecular response (EMR) (without T3151 mutation) | up to 6 months
  Time to achieve a response level (hematologic or molecular) is defined as the time from the date of the first dose of study treatment to the first documented achievement of each defined response level. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Time to achieve mplecular response (MR2) (without T3151 mutation) | up to 6 months
  Time to achieve a response level (hematologic or molecular) is defined as the time from the date of the first dose of study treatment to the first documented achievement of each defined response level. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Time to achieve major molecular response (MMR) (without T3151 mutation) | up to 6 months
  Time to achieve a response level (hematologic or molecular) is defined as the time from the date of the first dose of study treatment to the first documented achievement of each defined response level. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Time to achieve MR4 and MR4.5 (without T3151 mutation) | up to 6 months
  Time to achieve a response level (hematologic or molecular) is defined as the time from the date of the first dose of study treatment to the first documented achievement of each defined response level. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Duration of CHR (without T3151 mutation) | up to 6 months
  Duration of Response (DOR) is the time from the date of the first documented hematologic or molecular response level to the date of the first documented loss of the response level or death due to any cause, whichever occurs first. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Duration of EMR (without T3151 mutation) | up to 6 months
  Duration of Response (DOR) is the time from the date of the first documented hematologic or molecular response level to the date of the first documented loss of the response level or death due to any cause, whichever occurs first. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Duration of MR2 (without T3151 mutation) | up to 6 months
  Duration of Response (DOR) is the time from the date of the first documented hematologic or molecular response level to the date of the first documented loss of the response level or death due to any cause, whichever occurs first. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Duration of MMR (without T3151 mutation) | up to 6 months
  Duration of Response (DOR) is the time from the date of the first documented hematologic or molecular response level to the date of the first documented loss of the response level or death due to any cause, whichever occurs first. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Duration of MR4 & MR4.5 (without T3151 mutation) | up to 6 months
  Duration of Response (DOR) is the time from the date of the first documented hematologic or molecular response level to the date of the first documented loss of the response level or death due to any cause, whichever occurs first. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Percentage of participants with dose interruptions, reductions, and discontinuation (with T315I mutation) | up to 6 months
  Percentage of participants with dose interruptions, reductions, and discontinuation up to 6 months.
Percentage of participants achieving a CHR at 3 and 6 months of the treatment period (with T315I mutation) | up to 6 months
  A CHR is defined as the presence of all of the following for ≥4 weeks: white blood count (WBC) <10 x 109/L, platelet count <450 x 109/L, basophils <5%, no blasts and promyelocytes in peripheral blood, myelocytes + metamyelocytes <5% in peripheral blood, no evidence of extramedullary disease, including spleen and liver.
Percentage of participants achieving EMR at 3 and 6 months of the treatment period (with T315I mutation) | up to 6 months
  Levels of BCR::ABL1 transcripts will be determined by RQ-PCR testing of peripheral blood and analyzed at a central testing laboratory. Log reduction in BCR::ABL1 transcripts levels from the standardized baseline value, or the percent ratio of BCR::ABL1 transcripts versus control gene (ABL1) transcripts converted to a reference standard, will be calculated for each sample.
  Early molecular response (EMR) is defined as ≤10% BCR::ABL1 international scale (IS).
Percentage of participants achieving MR2 at 3 and 6 months of the treatment period (with T315I mutation) | up to 6 months
  Levels of BCR::ABL1 transcripts will be determined by RQ-PCR testing of peripheral blood and analyzed at a central testing laboratory. Log reduction in BCR::ABL1 transcripts levels from the standardized baseline value, or the percent ratio of BCR::ABL1 transcripts versus control gene (ABL1) transcripts converted to a reference standard, will be calculated for each sample. The rate of MR2 is defined as ≥2 log reduction of BCR::ABL (transcript from standardized baseline or ≤1% BCR::ABL/ABL1 % by IS), measured by RQ-PCR.
Percentage of participants achieving MMR at 3 and 6 months of the treatment period (with T315I mutation) | up to 6 months
  Levels of BCR::ABL1 transcripts will be determined by RQ-PCR testing of peripheral blood and analyzed at a central testing laboratory. Log reduction in BCR::ABL1 transcripts levels from the standardized baseline value, or the percent ratio of BCR::ABL1 transcripts versus control gene (ABL1) transcripts converted to a reference standard, will be calculated for each sample. Major molecular response (MMR) is defined as ≤0.1% BCR::ABL1 on the IS.
Percentage of participants achieving MR4 and MR4.5 at 3 and 6 months of the treatment period (with T315I mutation) | up to 6 months
  Levels of BCR::ABL1 transcripts will be determined by RQ-PCR testing of peripheral blood and analyzed at a central testing laboratory. Log reduction in BCR::ABL1 transcripts levels from the standardized baseline value, or the percent ratio of BCR::ABL1 transcripts versus control gene (ABL1) transcripts converted to a reference standard, will be calculated for each sample.
  MR4 is defined ≤0.01% BCR::ABL1 on the IS. MR4.5 is defined as ≤0.0032% BCR::ABL1 on the IS.
Time to achieve CHR during the treatment period (with T315I mutation) | Up to 6 months
  Time to achieve a response level (hematologic or molecular) is defined as the time from the date of the first dose of study treatment to the first documented achievement of each defined response level. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Time to achieve EMR during the treatment period (with T315I mutation) | Up to 6 months
  Time to achieve a response level (hematologic or molecular) is defined as the time from the date of the first dose of study treatment to the first documented achievement of each defined response level. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Time to achieve MR2 during the treatment period (with T315I mutation) | Up to 6 months
  Time to achieve a response level (hematologic or molecular) is defined as the time from the date of the first dose of study treatment to the first documented achievement of each defined response level. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Time to achieve MMR during the treatment period (with T315I mutation) | Up to 6 months
  ime to achieve a response level (hematologic or molecular) is defined as the time from the date of the first dose of study treatment to the first documented achievement of each defined response level. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Time to achieve MR4 and MR4.5 during the treatment period (with T315I mutation) | Up to 6 months
  Time to achieve a response level (hematologic or molecular) is defined as the time from the date of the first dose of study treatment to the first documented achievement of each defined response level. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Duration of CHR during the treatment period (with T315I mutation) | Up to 6 months
  Duration of Response (DOR) is the time from the date of the first documented hematologic or molecular response level to the date of the first documented loss of the response level or death due to any cause, whichever occurs first. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Duration of EMR during the treatment period (with T315I mutation) | Up to 6 months
  Duration of Response (DOR) is the time from the date of the first documented hematologic or molecular response level to the date of the first documented loss of the response level or death due to any cause, whichever occurs first. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Duration of MR2 during the treatment period (with T315I mutation) | Up to 6 months
  Duration of Response (DOR) is the time from the date of the first documented hematologic or molecular response level to the date of the first documented loss of the response level or death due to any cause, whichever occurs first. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Duration of MMR during the treatment period (with T315I mutation) | Up to 6 months
  Duration of Response (DOR) is the time from the date of the first documented hematologic or molecular response level to the date of the first documented loss of the response level or death due to any cause, whichever occurs first. It will be calculated for the treatment duration ie, up to 6 months from baseline.
Duration of MR4 and MR4.5 during the treatment period (with T315I mutation) | Up to 6 months
  Duration of Response (DOR) is the time from the date of the first documented hematologic or molecular response level to the date of the first documented loss of the response level or death due to any cause, whichever occurs first. It will be calculated for the treatment duration ie, up to 6 months from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- India (9):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Bengaluru, Karnataka
  - Novartis Investigative Site, Trivandrum, Kerala
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Cuttack
  - Novartis Investigative Site, Guwahati

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com